CLINICAL TRIAL: NCT05419908
Title: Pilot/Phase IIa Trial to Investigate the Effect of ESN364 in Early Postmenopausal Women Suffering From Hot Flashes
Brief Title: Trial to Investigate the Effect of ESN364 in Early Postmenopausal Women Suffering From Hot Flashes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ogeda S.A. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESN364_HF_204; 2015-002578-20 (EudraCT Number)
Record Dates: First submitted 2022-06-06; First posted 2022-06-15 (Actual); Results first posted 2023-07-25 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Hot Flashes
Keywords: Hot flashes; ESN364; ASP2693; fezolinetant; menopause; postmenopausal
MeSH Terms: conditions — Hot Flashes | interventions — fezolinetant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fezolinetant (Experimental): Participants received 90 milligrams (mg) fezolinetant capsules orally, twice daily (BID) for a period of 12 weeks
  Interventions: Drug: Fezolinetant
- Placebo (Placebo Comparator): Participants received fezolinetant matching placebo capsules orally, BID for a period of 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fezolinetant — Oral Capsule
  Other Names: ESN364; ASP2693
  Arms: Fezolinetant
Drug: Placebo — Oral Capsule
  Arms: Placebo

SUMMARY:
The primary purpose of this study was to evaluate the effect of ESN364 on the severity and frequency of hot flashes in early postmenopausal women suffering from hot flashes, in terms of changes in weekly Hot Flash Score from baseline to Week 12.

This study also evaluated the effect of ESN364 on the severity and frequency of hot flashes at additional timepoints; hot flash interference on daily life, in terms of changes from baseline over time in Hot Flash Related Daily Interference Scale (HFRDIS); the effect of ESN364 on climacteric symptoms, in terms of changes from baseline over time in Leeds Sleep Evaluation Questionnaire (LSEQ), Greene Climacteric Scale (GCS), and Sheehan Disability Scale (SDS); pharmacodynamic (PD) effect; and safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous amenorrhea for at least 12 consecutive months; or spontaneous amenorrhea for at least 6 months with biochemical criteria of menopause (FSH >40 IU/L); or spontaneous amenorrhea for at least 3 months with biochemical/physical criteria of menopause (FSH >40 IU/L and E2 <0.21 nmol/); or having had bilateral oophorectomy at least 6 weeks prior to screening (with or without hysterectomy);
* At least 49 moderate or severe hot flashes or night sweats over a period of 7 consecutive days, as recorded in the daily diary during the screening period, with at least 4 of those days with 7 or more moderate or severe hot flashes per day;
* In good general health as determined on the basis of medical history and general physical examination performed at screening; hematology and chemistry parameters, pulse rate and/or blood pressure, and ECG within the reference range for the population studied, or showing no clinically relevant deviations;
* Negative urine test for selected drugs of abuse (amphetamines, tricyclic antidepressants, cannabinoids, cocaine, tetrahydrocannabinol, or opiates) at screening;
* Negative serology panel (including hepatitis B surface antigen [HBsAg], antihepatitis C virus [HCV] and human immunodeficiency virus (HIV) antibody screens);
* Negative urine pregnancy test at screening;

Exclusion Criteria:

* Use of a prohibited therapy or not willing to wash-out drugs considered prohibited therapies;
* History (in the past year) or presence of drug or alcohol abuse;
* Suicide attempt in the past 3 years;
* Previous or current history of a malignant tumor (except basal cell carcinoma);
* Active liver disease or jaundice, or out-of-range values of alanine aminotransferase (ALT) and aspartate aminotransferase (AST); or total bilirubin >1.3 times the upper limit of normal (ULN); or creatinine >1.5 times the ULN; or estimated glomerular filtration rate (eGFR) using the Modification of Diet in Renal Disease (MDRD) formula <60 mL/min/1.73 m2 at screening;
* Medical condition or chronic disease (including history of neurological [including cognitive], hepatic, renal, cardiovascular, gastrointestinal, pulmonary [e.g., moderate asthma], or endocrine disease) or malignancy that could confound interpretation of the study outcome;
* Any psychological disorder according to the criteria indicated in the Diagnostics and Statistical Manual of Mental Disorders (DSM, 4th edition) within one year prior to screening. Such disorders include but are not limited to current major depression, alcohol (more than 3 glasses of wine, beer, or equivalent/day) or substance abuse/dependence;
* Unsuited to participate in the study, based on findings observed during physical examination, vital sign assessment, or 12-lead ECG;
* History of severe allergy, hypersensitivity, or intolerance to drugs in general, including the study drug and any of its excipients;
* Presence or sequellae of gastrointestinal, liver, kidney or other conditions known to interfere with the absorption, distribution, metabolism, or excretion (ADME) mechanisms of drugs;
* Concurrent participation in another interventional study (or participation within 3 months prior to screening in this study);
* History of poor compliance in clinical studies;
* Unable or unwilling to complete the study procedures;
* Subject is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff or relative thereof who is directly involved in the conduct of the study.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2016-09-21 (Actual); Study Completion 2016-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — Ogeda S.A.
Locations (8):
- Belgium (8):
  - Site BE32004, Brussels
  - Site BE32003, Genk
  - Site BE32001, Ghent
  - Site BE32006, Jette
  - Site BE32005, Kraainem
  - Site BE32007, Leuven
  - Site BE32008, Mons
  - Site BE32009, Tienen

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Result] Depypere H, Timmerman D, Donders G, Sieprath P, Ramael S, Combalbert J, Hoveyda HR, Fraser GL. Treatment of Menopausal Vasomotor Symptoms With Fezolinetant, a Neurokinin 3 Receptor Antagonist: A Phase 2a Trial. J Clin Endocrinol Metab. 2019 Dec 1;104(12):5893-5905. doi: 10.1210/jc.2019-00677. PMID 31415087
- See also: Link to plain language summary of the study on the Trial Results Summaries website. — http://www.trialsummaries.com/Study/StudyDetails?id=25137&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal women participants between 40 to 65 years of age who had hot flashes (HF) and who met the inclusion criteria and none of the exclusion criteria were enrolled in this study.
Pre-assignment Details: Prior to randomization, participants had a screening period during which a minimum 7-day collection of baseline HF frequency and severity assessments were performed.
Groups:
- Placebo: Participants received fezolinetant matching placebo capsules orally, twice daily (BID) for a period of 12 weeks.
- Fezolinetant: Participants received 90 milligrams (mg) fezolinetant capsules orally, BID for a period of 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Fezolinetant
Started | 44 | 43
Completed | 40 | 40
Not Completed | 4 | 3
Not completed — Participant Did not Fulfill all Inclusion/Exclusion Criteria | 1 | 0
Not completed — Serious Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Miscellaneous | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population was defined as all participants who were randomized into the study and received at least one dose of the study medication.
Groups:
- Fezolinetant: Participants received 90 mg fezolinetant capsules orally, BID for a period of 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Fezolinetant | Total
Number analyzed (Participants) | 44 | 43 | 87
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.7 (4.25) | 53.3 (4.03) | 53.5 (4.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 43 | 87
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 42 | 42 | 84
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 44 | 42 | 86
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Weekly General Hot Flash Score [Mean (Standard Deviation); unit: Score on a scale] — The HF Score was calculated as follows (number of mild HF/day × 1) + (number of moderate HF/day × 2) + (number of severe HF/day × 3). Higher scores indicate worse symptoms. There is no maximum score since the score was participant-dependent for both number and severity.
  Score on a scale | 25.76 (10.26) | 28.76 (13.39) | 27.24 (11.93)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in The Weekly General Hot Flash Score
Description: The HF score (based on severity and frequency) was calculated as:
  (number of mild HF/day × 1) + (number of moderate HF/day × 2) + (number of severe HF/day × 3)
  The severity of HFs is clinically defined as follows:
  * Mild: sensation of heat without sweating/dampness. If at night, participant didn't wake up but later notices damp sheets or clothing.
  * Moderate: Sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets.
  * Severe: Sensation of intense heat with sweating, causing disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., removing layers of clothes, open the window, or get out of bed).
  Higher scores indicate worse symptoms. There is no maximum score since the score was participant dependent for both number and severity.
Time Frame: Baseline and week 12
Population: Intent-to-treat (ITT) population (included all randomized participants who received at least one dose of the study medication and who had post-baseline efficacy data) with available data at specified time point.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 40 | 40
score on a scale | -12.19 [-16.55 to -7.83] | -26.51 [-30.83 to -22.18]
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant; Test type: Superiority; p < 0.001, ANCOVA — Least square (LS) mean difference versus placebo, obtained from an ANCOVA model with treatment group as fixed effect and baseline weekly hot flash score as covariate. P-value of the t-statistic testing whether there is a treatment difference; Analysis of Covariance (ANCOVA); LSMean Difference = -12.34, 95% CI 2-sided [-16.89 to -7.79]

2. Secondary Outcome: Change From Baseline in The Weekly Hot Flash Severity Score at Weeks 4, 8 and 12 (Method 1)
Description: The HF Severity Score by method 1 takes into account the number and severity of moderate and severe HF occurred during a given time period and was calculated as follows HF Severity score = [(number of moderate HF/day × 2) + (number of severe HF/day × 3)]/(number of moderate HF + number of severe HF)
  The severity of HFs was clinically defined as follows:
  * Moderate: Sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets.
  * Severe: Sensation of intense heat with sweating, causing disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., removing layers of clothes, open the window, or get out of bed).
  Higher scores indicate worse symptoms. There is no maximum score since the score was participant-dependent for both number and severity.
Time Frame: Baseline and weeks 4, 8 and 12
Population: ITT population with available data at specified time point.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 44 | 41
score on a scale
  Week 4 | -0.294 [-0.473 to -0.116] | -1.428 [-1.718 to -1.138]
  Week 8: number analyzed (Participants) | 41 | 40
  Week 8 | -0.608 [-0.899 to -0.318] | -1.557 [-1.858 to -1.257]
  Week 12: number analyzed (Participants) | 40 | 40
  Week 12 | -0.534 [-0.798 to -0.270] | -1.656 [-1.937 to -1.376]
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant; Week 4; Test type: Superiority; p < 0.001, ANCOVA — Least square mean difference versus placebo, obtained from an ANCOVA model with treatment group as fixed effect and baseline weekly hot flash score as covariate. P-value of the t-statistic testing whether there is a treatment difference; LSMean Difference = -1.134, 95% CI 2-sided [-1.466 to -0.802]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant; Week 8; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LSMean Difference = -0.948, 95% CI [-1.362 to -0.535]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant; Week 12; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LSMean Difference = -1.122, 95% CI 2-sided [-1.504 to -0.741]

3. Secondary Outcome: Change From Baseline in The Weekly Hot Flash Severity Score at Weeks 4, 8 and 12 (Method 2)
Description: The HF Severity Score by method 2 takes into account moderate and severe HF during a given time period and was calculated as follows HF Severity score = [(number of moderate HF/day × 2) + (number of severe HF/day × 3)]
  The severity of HFs was clinically defined as follows:
  * Moderate: Sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets.
  * Severe: Sensation of intense heat with sweating, causing disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., removing layers of clothes, open the window, or get out of bed).
  Higher scores indicate worse symptoms. There is no maximum score since the score was participant-dependent for both number and severity.
Time Frame: Baseline and weeks 4, 8 and 12
Population: ITT population with available data at specified time point.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 44 | 41
score on a scale
  Week 4 | -9.55 [-12.73 to -6.36] | -25.26 [-29.64 to -20.89]
  Week 8: number analyzed (Participants) | 41 | 41
  Week 8 | -11.91 [-15.72 to -8.10] | -25.71 [-30.15 to -21.27]
  Week 12: number analyzed (Participants) | 40 | 40
  Week 12 | -12.14 [-16.62 to -7.65] | -26.61 [-31.06 to -22.17]
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant; Week 4; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LSMean Difference = -13.28, 95% CI [-17.02 to -9.54]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant; Week 8; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LSMean Difference = -11.78, 95% CI 2-sided [-16.30 to -7.27]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant; Week 12; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LSMean Difference = -12.42, 95% CI [-17.00 to -7.83]

4. Secondary Outcome: Change From Baseline in The Weekly Mild, Moderate and Severe Hot Flash Frequency at Weeks 4, 8 and 12
Description: The weekly HF frequency was calculated as number of mild, moderate and severe hot flashes over the week.
  * Mild: sensation of heat without sweating/dampness. If at night, participant didn't wake up but later notices damp sheets or clothing.
  * Moderate: Sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets.
  * Severe: Sensation of intense heat with sweating, causing disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., removing layers of clothes, open the window, or get out of bed).
  Higher number of hot flashes is worse.
Time Frame: Baseline and weeks 4, 8 and 12
Population: ITT population with available data at specified time point.
Measure: Mean (95% Confidence Interval); unit: HF's per day
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 44 | 41
HF's per day
  Week 4 | -26.4 [-35.2 to -17.5] | -72.3 [-82.7 to -61.8]
  Week 8: number analyzed (Participants) | 41 | 40
  Week 8 | -32.9 [-43.2 to -22.7] | -73.3 [-83.8 to -62.8]
  Week 12: number analyzed (Participants) | 40 | 40
  Week 12 | -35.6 [-46.7 to -24.5] | -75.3 [-86.4 to -64.3]
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant; Week 4; Test type: Superiority; p < 0.001, ANCOVA — Least square mean difference versus placebo, obtained from an ANCOVA model with treatment group as factor. P-value of the t-statistic testing whether there is a treatment difference; LSMean Difference = -39.8, 95% CI 2-sided [-50.5 to -29.1]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant; Week 8; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LSMean Difference = -35.5, 95% CI 2-sided [-47.9 to -23.0]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant; Week 12; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LSMean Difference = -35.0, 95% CI [-47.9 to -22.1]

5. Secondary Outcome: Percentage of Participants With >=70% Reduction in the Weekly Hot Flash Score From Baseline to Weeks 4, 8 and 12
Description: The HF score (based on severity and frequency) was calculated as:
  (number of mild HF/day × 1) + (number of moderate HF/day × 2) + (number of severe HF/day × 3)
  The severity of HFs is clinically defined as follows:
  * Mild: sensation of heat without sweating/dampness. If at night, participant didn't wake up but later notices damp sheets or clothing.
  * Moderate: Sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets.
  * Severe: Sensation of intense heat with sweating, causing disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., removing layers of clothes, open the window, or get out of bed).
  Higher scores indicate worse symptoms. There is no maximum score since the score was participant-dependent for both number and severity.
Time Frame: Baseline and weeks 4, 8 and 12
Population: ITT population with available data at specified time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 44 | 41
percentage of participants
  Week 4 | 22.7 [10.34 to 35.11] | 87.8 [77.79 to 97.82]
  Week 8: number analyzed (Participants) | 41 | 40
  Week 8 | 39.0 [24.09 to 53.96] | 87.5 [77.25 to 97.75]
  Week 12: number analyzed (Participants) | 40 | 40
  Week 12 | 42.5 [27.18 to 57.82] | 95.0 [88.25 to 100.00]
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant; Week 4; Test type: Superiority; p < 0.001, Likelihood-Ratio Chi-Square Test — Likelihood-ratio test based 95% confidence interval of the percentage difference; Percentage Difference = 65.1, 95% CI 2-sided [49.15 to 81.00]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant; Week 8; Test type: Superiority; p < 0.001, Likelihood-Ratio Chi-Square Test — Likelihood-ratio test based 95% confidence interval of the percentage difference; Percentage Difference = 48.5, 95% CI [30.37 to 66.59]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant; Week 12; Test type: Superiority; p < 0.001, Likelihood-Ratio Chi-Square Test — Likelihood-ratio test based 95% confidence interval of the percentage difference; Percentage Difference = 52.5, 95% CI 2-sided [35.76 to 69.24]

6. Secondary Outcome: Percentage of Participants With >=80% Reduction in the Weekly Hot Flash Score From Baseline to Weeks 4, 8 and 12
Description: as for outcome 5
Time Frame: Baseline and weeks 4, 8 and 12
Population: ITT population with available data at specified time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 44 | 41
percentage of participants
  Week 4 | 9.1 [0.60 to 17.59] | 78.0 [65.38 to 90.72]
  Week 8: number analyzed (Participants) | 41 | 40
  Week 8 | 26.8 [13.27 to 40.39] | 77.5 [64.56 to 90.44]
  Week 12: number analyzed (Participants) | 40 | 40
  Week 12 | 30.0 [15.80 to 44.20] | 87.5 [77.25 to 97.75]
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant; Week 4; Test type: Superiority; p < 0.001, Likelihood-Ratio Chi-Square Test — Likelihood-ratio test based 95% confidence interval of the percentage difference; Percentage Difference = 69.0, 95% CI 2-sided [53.70 to 84.21]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant; Week 8; Test type: Superiority; p < 0.001, Likelihood-Ratio Chi-Square Test — Likelihood-ratio test based 95% confidence interval of the percentage difference; Percentage Difference = 50.7, 95% CI [31.93 to 69.42]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant; Week 12; Test type: Superiority; p < 0.001, Likelihood-Ratio Chi-Square Test — Likelihood-ratio test based 95% confidence interval of the percentage difference; Percentage Difference = 57.5, 95% CI 2-sided [39.99 to 75.01]

7. Secondary Outcome: Percentage of Participants With >=90% Reduction in the Weekly Hot Flash Score From Baseline to Weeks 4, 8 and 12
Description: The HF score (based on severity and frequency) was calculated as:
  (number of mild HF/day × 1) + (number of moderate HF/day × 2) + (number of severe HF/day × 3)
  The severity of HF is clinically defined as follows:
  * Mild: sensation of heat without sweating/dampness. If at night, participant didn't wake up but later notices damp sheets or clothing.
  * Moderate: Sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets.
  * Severe: Sensation of intense heat with sweating, causing disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., removing layers of clothes, open the window, or get out of bed).
  Higher scores indicate worse symptoms. There is no maximum score since the score was participant-dependent for both number and severity.
Time Frame: Baseline and weeks 4, 8 and 12
Population: ITT population with available data at specified time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 44 | 41
percentage of participants
  Week 4 | 6.8 [0.00 to 14.27] | 61.0 [46.04 to 75.91]
  Week 8: number analyzed (Participants) | 41 | 40
  Week 8 | 12.2 [2.18 to 22.21] | 60.0 [44.82 to 75.18]
  Week 12: number analyzed (Participants) | 40 | 40
  Week 12 | 15.0 [3.93 to 26.07] | 62.5 [47.50 to 77.50]
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant; Week 4; Test type: Superiority; p < 0.001, Likelihood-Ratio Chi-Square Test — Likelihood-ratio test based 95% confidence interval of the percentage difference; Percentage Difference = 54.2, 95% CI 2-sided [37.47 to 70.84]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant; Week 8; Test type: Superiority; p < 0.001, Likelihood-Ratio Chi-Square Test — Likelihood-ratio test based 95% confidence interval of the percentage difference; Percentage Difference = 47.8, 95% CI [29.62 to 65.99]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant; Week 12; Test type: Superiority; p < 0.001, Likelihood-Ratio Chi-Square Test — Likelihood-ratio test based 95% confidence interval of the percentage difference; Percentage Difference = 47.5, 95% CI [28.86 to 66.14]

8. Secondary Outcome: Percentage of Participants With >=50% Reduction in the Weekly Frequency of Moderate and Severe HF From Baseline to Weeks 4, 8 and 12
Description: The weekly HF frequency of moderate and severe HF was calculated as number of moderate and severe HF over the week.
  * Moderate: Sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets.
  * Severe: Sensation of intense heat with sweating, causing disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., removing layers of clothes, open the window, or get out of bed).
  Higher number of HF indicates worse symptoms.
Time Frame: Baseline and weeks 4, 8 and 12
Population: ITT population with available data at specified time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 44 | 41
percentage of participants
  Week 4 | 45.5 [30.74 to 60.17] | 95.1 [88.53 to 100.00]
  Week 8: number analyzed (Participants) | 41 | 40
  Week 8 | 53.7 [38.39 to 68.92] | 97.5 [92.66 to 100.00]
  Week 12: number analyzed (Participants) | 40 | 40
  Week 12 | 55.0 [39.58 to 70.42] | 97.5 [92.66 to 100.00]
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant; Week 4; Test type: Superiority; p < 0.001, Likelihood-Ratio Chi-Square Test — Likelihood-ratio test based 95% confidence interval of the percentage difference; Percentage Difference = 49.7, 95% CI [33.54 to 65.79]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant; Week 8; Test type: Superiority; p < 0.001, Likelihood-Ratio Chi-Square Test — Likelihood-ratio test based 95% confidence interval of the percentage difference; Percentage Difference = 43.8, 95% CI 2-sided [27.83 to 59.85]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant; Week 12; Test type: Superiority; p < 0.001, Likelihood-Ratio Chi-Square Test — Likelihood-ratio test based 95% confidence interval of the percentage difference; Percentage Difference = 42.5, 95% CI [26.34 to 58.66]

9. Secondary Outcome: Percentage of Participants With >=70% Reduction in the Weekly Frequency of Moderate and Severe HF From Baseline to Weeks 4, 8 and 12
Description: as for outcome 8
Time Frame: Baseline and weeks 4, 8 and 12
Population: ITT population with available data at specified time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 44 | 41
percentage of participants
  Week 4 | 25.0 [12.21 to 37.79] | 87.8 [77.79 to 97.82]
  Week 8: number analyzed (Participants) | 41 | 40
  Week 8 | 46.3 [31.08 to 61.61] | 92.5 [84.34 to 100.00]
  Week 12: number analyzed (Participants) | 40 | 40
  Week 12 | 40.0 [24.82 to 55.18] | 97.5 [92.66 to 100.00]
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant; Week 4; Test type: Superiority; p < 0.001, Likelihood-Ratio Chi-Square Test — Likelihood-ratio test based 95% confidence interval of the percentage difference; Percentage Difference = 62.8, 95% CI 2-sided [46.56 to 79.05]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant; Week 8; Test type: Superiority; p < 0.001, Likelihood-Ratio Chi-Square Test — Likelihood-ratio test based 95% confidence interval of the percentage difference; Percentage Difference = 46.2, 95% CI 2-sided [28.85 to 63.47]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant; Week 12; Test type: Superiority; p < 0.001, Likelihood-Ratio Chi-Square Test — Likelihood-ratio test based 95% confidence interval of the percentage difference; Percentage Difference = 57.5, 95% CI 2-sided [41.57 to 73.43]

10. Secondary Outcome: Percentage of Participants With >=90% Reduction in the Weekly Frequency of Moderate and Severe HF From Baseline to Weeks 4, 8 and 12
Description: as for outcome 8
Time Frame: Baseline and weeks 4, 8 and 12
Population: ITT population with available data at specified time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 44 | 41
percentage of participants
  Week 4 | 6.8 [0.00 to 14.27] | 68.3 [54.05 to 82.54]
  Week 8: number analyzed (Participants) | 41 | 40
  Week 8 | 24.4 [11.25 to 37.54] | 67.5 [52.99 to 82.01]
  Week 12: number analyzed (Participants) | 40 | 40
  Week 12 | 20.0 [7.60 to 32.40] | 72.5 [58.66 to 86.34]
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant; Week 4; Test type: Superiority; p < 0.001, Likelihood-Ratio Chi-Square Test — Likelihood-ratio test based 95% confidence interval of the percentage difference; Percentage Difference = 61.5, 95% CI [45.40 to 77.55]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant; Week 8; Test type: Superiority; p < 0.001, Likelihood-Ratio Chi-Square Test — Likelihood-ratio test based 95% confidence interval of the percentage difference; Percentage Difference = 43.1, 95% CI 2-sided [23.53 to 62.69]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant; Week 12; Test type: Superiority; p < 0.001, Likelihood-Ratio Chi-Square Test — Likelihood-ratio test based 95% confidence interval of the percentage difference; Percentage Difference = 52.5, 95% CI [33.92 to 71.08]

11. Secondary Outcome: Change From Baseline in Hot Flash Related Daily Interference Scale (HFRDIS) Score at Weeks 4, 8 and 12
Description: The HFRDIS was a 10-item scale which measured a woman's perceptions of the degree to which HF interfere with 9 daily life activities (work, social activities, leisure, sleep, mood, concentration, relations with others, sexuality, enjoying life); the 10th item measures interference with overall quality of life. This scale was modeled after items on the Brief Pain Inventory and Brief Fatigue Inventory both of which assessed the extent to which pain or fatigue interfere with daily life. Participants were asked to rate the extent to which HF had interfered with each item during the previous 4-week time interval using a 0 (do not interfere) to 10 (completely interfere) scale. Overall mean score was calculated as sum of items/number of available items. Higher score indicate a higher interference.
Time Frame: Baseline and weeks 4, 8 and 12
Population: ITT population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 42 | 41
score on a scale
  Week 4: Work | -1.7 (2.93) | -4.6 (2.65)
  Week 8: Work: number analyzed (Participants) | 39 | 39
  Week 8: Work | -2.4 (2.80) | -5.0 (2.38)
  Week 12: Work: number analyzed (Participants) | 39 | 39
  Week 12: Work | -2.3 (2.58) | -4.6 (2.68)
  Week 4: Social Activities | -1.6 (2.53) | -4.3 (2.48)
  Week 8: Social Activities: number analyzed (Participants) | 39 | 39
  Week 8: Social Activities | -1.9 (2.85) | -4.7 (2.37)
  Week 12: Social Activities: number analyzed (Participants) | 39 | 39
  Week 12: Social Activities | -1.8 (2.51) | -4.3 (2.35)
  Week 4: Leisure Activities | -1.6 (2.63) | -4.0 (2.51)
  Week 8: Leisure Activities: number analyzed (Participants) | 39 | 39
  Week 8: Leisure Activities | -1.7 (2.72) | -4.2 (2.50)
  Week 12: Leisure Activities: number analyzed (Participants) | 39 | 39
  Week 12: Leisure Activities | -2.0 (2.52) | -3.8 (3.08)
  Week 4: Sleep | -2.5 (2.93) | -5.2 (2.77)
  Week 8: Sleep: number analyzed (Participants) | 39 | 39
  Week 8: Sleep | -3.2 (3.29) | -5.7 (2.37)
  Week 12: Sleep: number analyzed (Participants) | 39 | 39
  Week 12: Sleep | -3.3 (3.01) | -5.8 (2.43)
  Week 4: Mood | -2.3 (2.49) | -4.0 (2.85)
  Week 8: Mood: number analyzed (Participants) | 39 | 39
  Week 8: Mood | -2.3 (2.86) | -4.4 (2.84)
  Week 12: Mood: number analyzed (Participants) | 39 | 39
  Week 12: Mood | -2.5 (2.56) | -4.3 (2.64)
  Week 4: Concentration | -1.6 (2.68) | -3.9 (2.57)
  Week 8: Concentration: number analyzed (Participants) | 39 | 39
  Week 8: Concentration | -1.6 (3.06) | -4.1 (2.59)
  Week 12: Concentration: number analyzed (Participants) | 39 | 39
  Week 12: Concentration | -1.9 (3.17) | -4.0 (2.47)
  Week 4: Relations With Others | -2.1 (2.93) | -3.3 (2.45)
  Week 8: Relations With Others: number analyzed (Participants) | 39 | 39
  Week 8: Relations With Others | -1.8 (3.02) | -3.5 (2.70)
  Week 12: Relations With Others: number analyzed (Participants) | 39 | 39
  Week 12: Relations With Others | -1.8 (3.16) | -3.3 (2.67)
  Week 4: Sexuality | -1.9 (2.88) | -3.0 (3.49)
  Week 8: Sexuality: number analyzed (Participants) | 39 | 39
  Week 8: Sexuality | -1.8 (3.48) | -3.2 (3.76)
  Week 12: Sexuality: number analyzed (Participants) | 39 | 39
  Week 12: Sexuality | -1.7 (2.84) | -3.4 (3.86)
  Week 4: Enjoyment of Life | -1.6 (2.86) | -3.6 (2.65)
  Week 8: Enjoyment of Life: number analyzed (Participants) | 39 | 39
  Week 8: Enjoyment of Life | -1.5 (3.15) | -3.9 (2.59)
  Week 12: Enjoyment of Life: number analyzed (Participants) | 39 | 39
  Week 12: Enjoyment of Life | -1.6 (3.38) | -3.7 (2.42)
  Week 4: Overall Quality of Life | -1.4 (2.43) | -3.8 (2.87)
  Week 8: Overall Quality of Life: number analyzed (Participants) | 39 | 39
  Week 8: Overall Quality of Life | -1.5 (3.01) | -4.5 (1.92)
  Week 12: Overall Quality of Life: number analyzed (Participants) | 39 | 39
  Week 12: Overall Quality of Life | -1.6 (3.05) | -4.6 (2.16)
  Week 4: Overall Mean Score | -1.84 (1.922) | -3.97 (2.141)
  Week 8: Overall Mean Score: number analyzed (Participants) | 39 | 39
  Week 8: Overall Mean Score | -1.98 (2.439) | -4.33 (1.945)
  Week 12: Overall Mean Score: number analyzed (Participants) | 39 | 39
  Week 12: Overall Mean Score | -2.05 (2.326) | -4.17 (2.067)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant; Week 4: Work; Test type: Superiority; p < 0.001, ANCOVA — Least square mean difference versus placebo, obtained from an ANCOVA model with treatment group as fixed effect and baseline weekly hfrdis as covariate; LSMean Difference = -2.53, 95% CI 2-sided [-3.45 to -1.60]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant; Week 8: Work; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -2.29, 95% CI 2-sided [-3.15 to -1.42]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant; Week 12: Work; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -2.11, 95% CI 2-sided [-3.03 to -1.20]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant; Week 4: Social Activities; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -2.33, 95% CI 2-sided [-3.19 to -1.46]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant; Week 8: Social Activties; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -2.34, 95% CI 2-sided [-3.21 to -1.47]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant; Week 12: Social Activties; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -2.19, 95% CI 2-sided [-3.09 to -1.29]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant; Week 4: Leisure Activities; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -2.15, 95% CI 2-sided [-2.99 to -1.31]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant; Week 8: Leisure Activties; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -2.37, 95% CI 2-sided [-3.19 to -1.55]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant; Week 12: Leisure Activties; Test type: Superiority; p = 0.002, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -1.64, 95% CI 2-sided [-2.66 to -0.62]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant; Week 4: Sleep; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -2.93, 95% CI 2-sided [-4.08 to -1.78]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant; Week 8: Sleep; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -2.71, 95% CI 2-sided [-3.86 to -1.57]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant; Week 12: Sleep; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -2.61, 95% CI 2-sided [-3.67 to -1.54]
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant; Week 4: Mood; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -1.74, 95% CI 2-sided [-2.67 to -0.81]
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant; Week 8: Mood; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -2.12, 95% CI 2-sided [-3.09 to -1.16]
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant; Week 12: Mood; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -1.79, 95% CI 2-sided [-2.69 to -0.88]
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant; Week 4: Concentration; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -1.92, 95% CI 2-sided [-2.86 to -0.97]
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant; Week 8: Concentration; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -2.23, 94% CI 2-sided [-3.21 to -1.25]
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant; Week 12: Concentration; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -1.90, 95% CI 2-sided [-2.91 to -0.88]
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant; Week 4: Relations With Others; Test type: Superiority; p = 0.003, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -1.33, 95% CI 2-sided [-2.20 to -0.46]
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant; Week 8: Relations With others; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -1.85, 95% CI 2-sided [-2.80 to -0.90]
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant; Week 12: Relations With Others; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -1.72, 95% CI 2-sided [-2.66 to -0.77]
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant; Week 4: Sexuality; Test type: Superiority; p = 0.081, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -1.06, 95% CI 2-sided [-2.25 to 0.13]
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant; Week 8: Sexuality; Test type: Superiority; p = 0.050, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -1.40, 95% CI 2-sided [-2.80 to 0.00]
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant; Week 12: Sexuality; Test type: Superiority; p = 0.026, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -1.51, 95% CI 2-sided [-2.84 to -0.19]
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant; Week 4: Enjoyment of Life; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -1.65, 95% CI 2-sided [-2.51 to -0.79]
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant; Week 8: Enjoyment of Life; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -2.07, 95% CI 2-sided [-2.97 to -1.18]
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant; Week 12: Enjoyment of Life; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -1.83, 95% CI 2-sided [-2.88 to -0.78]
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant; Week4: Overall Quality of Life; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean difference = -1.92, 95% CI 2-sided [-2.86 to -0.97]
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant; Week 8: Overall Quality of Life; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -2.51, 95% CI 2-sided [-3.41 to -1.61]
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant; Week 12: Overall Quality of Life; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -2.36, 95% CI 2-sided [-3.31 to -1.41]
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant; Week 4: Overall Mean Score; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -1.98, 95% CI 2-sided [-2.73 to -1.23]
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant; Week 8: Overall Mean Score; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -2.21, 95% CI 2-sided [-3.02 to -1.40]
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant; Week 12: Overall Mean Score; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 11, analysis 1]; LSMean Difference = -1.98, 95% CI 2-sided [-2.83 to -1.13]

12. Secondary Outcome: Change From Baseline in Leeds Sleep Evaluation Questionnaire (LSEQ) at Weeks 4, 8 and 12
Description: The LSEQ was a 10-item self-rated questionnaire which assessed participants aspects of sleep and early morning behavior. The questions were grouped into 4 chronological areas: the ease of getting to sleep, the perceived quality of sleep, the ease of awaking from sleep, and the integrity of early morning behavior following wakefulness. The LSEQ was a visual analogue scale which requires respondents to place marks on a group of 10 cm lines. representing the changes they have experienced in a variety of symptoms since the beginning of treatment. Lines extends between extremes like "more difficult than usual" and "easier than usual". Responses are measured using a 100-mm scale and are averaged to provide a score for each domain.
Time Frame: Baseline and weeks 4, 8 and 12
Population: ITT population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 43 | 41
millimeter (mm)
  Week 4: Getting to Sleep | 1.017 (1.9195) | 2.283 (2.7364)
  Week 8: Getting to Sleep: number analyzed (Participants) | 40 | 40
  Week 8: Getting to Sleep | 1.145 (1.7931) | 2.248 (2.5233)
  Week 12: Getting to Sleep: number analyzed (Participants) | 39 | 39
  Week 12: Getting to Sleep | 1.282 (1.7761) | 2.094 (2.4419)
  Week 4: Quality of Sleep | 2.145 (2.6443) | 4.437 (4.0768)
  Week 8: Quality of Sleep: number analyzed (Participants) | 39 | 40
  Week 8: Quality of Sleep | 2.378 (2.8160) | 4.703 (3.1971)
  Week 12: Quality of Sleep: number analyzed (Participants) | 39 | 39
  Week 12: Quality of Sleep | 1.904 (2.7872) | 4.385 (3.4477)
  Week 4: Awake Following Sleep: number analyzed (Participants) | 43 | 40
  Week 4: Awake Following Sleep | 0.642 (2.0739) | 2.180 (3.0579)
  Week 8: Awake Following Sleep: number analyzed (Participants) | 40 | 40
  Week 8: Awake Following Sleep | 0.653 (2.5019) | 2.920 (3.0219)
  Week 12: Awake Following Sleep: number analyzed (Participants) | 39 | 39
  Week 12: Awake Following Sleep | 1.024 (2.6114) | 2.887 (3.1333)
  Week 4: Behavior Following Wakening | 1.173 (2.1743) | 2.513 (2.7919)
  Week 8: Behavior Following Wakening: number analyzed (Participants) | 40 | 40
  Week 8: Behavior Following Wakening | 0.750 (2.6371) | 2.539 (2.7742)
  Week 12: Behavior Following Wakening: number analyzed (Participants) | 39 | 39
  Week 12: Behavior Following Wakening | 1.203 (2.5185) | 2.233 (2.8190)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant; Week 4: Getting to Sleep; Test type: Superiority; p < 0.001, ANCOVA — Least square mean difference versus placebo, obtained from an ANCOVA model with treatment group as fixed effect and baseline LSEQ as covariate; LSMean Difference = 1.375, 95% CI 2-sided [0.651 to 2.100]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant; Week 8: Getting to Sleep; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; LSMean Difference = 1.166, 95% CI 2-sided [0.505 to 1.827]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant; Week 12: Getting to Sleep; Test type: Superiority; p = 0.014, ANCOVA — [p-value comment as in outcome 12, analysis 1]; LSMean Difference = 0.895, 95% CI 2-sided [0.190 to 1.599]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant; Week 4: Quality of Sleep; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; LSMean Difference = 2.423, 95% CI 2-sided [1.308 to 3.539]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant; Week 8: Quality of Sleep; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; LSMean Difference = 2.291, 95% CI 2-sided [1.31 to 3.251]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant; Week 12: Quality of Sleep; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; LSMean Difference = 2.433, 95% CI 2-sided [1.334 to 3.532]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant; Week 4: Awake Following Sleep; Test type: Superiority; p = 0.059, ANCOVA — [p-value comment as in outcome 12, analysis 1]; LSMean Difference = 0.877, 95% CI 2-sided [-0.034 to 1.789]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant; Week 8: Awake Following Sleep; Test type: Superiority; p = 0.001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; LSMean Difference = 1.457, 95% CI 2-sided [0.579 to 2.335]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant; Week 12: Awake Following Sleep; Test type: Superiority; p = 0.031, ANCOVA — [p-value comment as in outcome 12, analysis 1]; LSMean Difference = 1.113, 95% CI 2-sided [0.107 to 2.120]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant; Week 4: Behaviour Following Wakening; Test type: Superiority; p = 0.008, ANCOVA — [p-value comment as in outcome 12, analysis 1]; LSMean Difference = 1.203, 95% CI 2-sided [0.317 to 2.088]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant; Week 8: Behaviour Following Wakening; Test type: Superiority; p = 0.001, ANCOVA — [p-value comment as in outcome 12, analysis 1]; LSMean Difference = 1.597, 95% CI 2-sided [0.639 to 2.556]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant; Week 12: Behaviour Following Sleep; Test type: Superiority; p = 0.084, ANCOVA — [p-value comment as in outcome 12, analysis 1]; LSMean Difference = 0.842, 95% CI 2-sided [-0.116 to 1.800]

13. Secondary Outcome: Change From Baseline in Greene Climacteric Scale (GCS) at Weeks 4, 8 and 12
Description: The GCS was a 21-item scale which provides a brief but comprehensive and valid measure of climacteric symptomatology. Each item was rated by the participant according to its severity using a four-point rating scale from 0 (none) to 3 (severe). The first 20 items of the scale combine into three main independent symptom measures: psychological symptoms (items 1 to 11; score 0 to 33), physical symptoms (items 12 to 18; score 0 to 21), and vasomotor symptoms (items 19 to 20; score 0 to 6), by summing up the individual item scores. Item 21 is a probe for sexual dysfunction (Loss of interest in sex). The total score ranges from 0 to 63. Higher scores indicate worse symptoms.
Time Frame: Baseline and weeks 4, 8 and 12
Population: ITT population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 43 | 40
score on a scale
  Week 4: Loss of Interest in Sex: number analyzed (Participants) | 41 | 40
  Week 4: Loss of Interest in Sex | -0.4 (0.67) | -0.5 (0.88)
  Week 8: Loss of interest in Sex: number analyzed (Participants) | 39 | 39
  Week 8: Loss of interest in Sex | -0.5 (0.85) | -0.7 (1.15)
  Week 12: Loss of Interest in Sex: number analyzed (Participants) | 39 | 39
  Week 12: Loss of Interest in Sex | -0.4 (0.75) | -0.6 (1.14)
  Week 4: Psychological: number analyzed (Participants) | 41 | 39
  Week 4: Psychological | -2.3 (5.22) | -5.3 (5.97)
  Week 8: Psychological: number analyzed (Participants) | 39 | 38
  Week 8: Psychological | -2.6 (5.31) | -6.7 (6.49)
  Week 12: Psychological: number analyzed (Participants) | 38 | 39
  Week 12: Psychological | -2.9 (5.14) | -6.6 (6.03)
  Week 4: Physical: number analyzed (Participants) | 39 | 38
  Week 4: Physical | -2.1 (3.68) | -1.2 (2.71)
  Week 8: Physical: number analyzed (Participants) | 37 | 38
  Week 8: Physical | -1.9 (3.46) | -1.9 (3.09)
  Week 12: Physical: number analyzed (Participants) | 38 | 37
  Week 12: Physical | -2.4 (3.80) | -1.9 (3.32)
  Week 4: Vasomotor | -1.1 (1.79) | -3.3 (1.83)
  Week 8: Vasomotor: number analyzed (Participants) | 39 | 39
  Week 8: Vasomotor | -1.7 (2.23) | -3.6 (1.48)
  Week 12: Vasomotor: number analyzed (Participants) | 40 | 39
  Week 12: Vasomotor | -1.5 (2.31) | -3.6 (1.37)
  Week 4: Total Symptom Score: number analyzed (Participants) | 37 | 35
  Week 4: Total Symptom Score | -5.5 (9.33) | -9.9 (9.24)
  Week 8: Total Symptom Score: number analyzed (Participants) | 34 | 35
  Week 8: Total Symptom Score | -5.8 (8.89) | -13.1 (10.68)
  Week 12: Total Symptom Score: number analyzed (Participants) | 36 | 35
  Week 12: Total Symptom Score | -6.3 (8.87) | -13.1 (10.04)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant; Week 4: Loss of Interest in Sex; Test type: Superiority; p = 0.881, ANCOVA — Least square mean difference versus placebo, obtained from an ANCOVA model with treatment group as fixed effect and baseline GCS as covariate; LSMean Difference = 0.00, 95% CI 2-sided [-0.3 to 0.3]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant; Week 8: Loss of Interest in Sex; Test type: Superiority; p = 0.383, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LSMean Difference = -0.2, 95% CI 2-sided [-0.6 to 0.2]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant; Week 12: Loss of Interest in Sex; Test type: Superiority; p = 0.301, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LSMean Difference = -0.2, 95% CI 2-sided [-0.6 to 0.2]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant; Week 4: Psychological; Test type: Superiority; p = 0.020, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LSMean Difference = -2.5, 95% CI 2-sided [-4.5 to -0.4]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant; Week 8: Psychological; Test type: Superiority; p = 0.003, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LSMean Difference = -3.3, 95% CI 2-sided [-5.4 to -1.2]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant; Week 12: Psychological; Test type: Superiority; p = 0.005, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LSMean Difference = -3.1, 95% CI 2-sided [-5.2 to -1.0]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant; Week 4: Physical; Test type: Superiority; p = 0.732, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LSMean Difference = -0.2, 95% CI 2-sided [-1.2 to 0.9]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant; Week 8: Physical; Test type: Superiority; p = 0.282, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LSMean Difference = -0.7, 95% CI 2-sided [-1.9 to 0.6]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant; Week 12: Physical; Test type: Superiority; p = 0.254, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LSMean Difference = -0.6, 95% CI 2-sided [-1.7 to 0.5]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant; Week 4: Vasomotor; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LSMean Difference = -2.0, 95% CI 2-sided [-2.7 to -1.4]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant; Week 8: Vasomotor; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LSMean Difference = -1.8, 95% CI 2-sided [-2.4 to -1.1]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant; Week 12: Vasomotor; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LSMean Difference = -2.0, 95% CI 2-sided [-2.6 to -1.3]
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant; Week 4: Total Symptom Score; Test type: Superiority; p = 0.013, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LSMean Difference = -4.6, 95% CI 2-sided [-8.2 to -1.0]
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant; Week 8: Total Symptom Score; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LSMean Difference = -6.9, 95% CI 2-sided [-10.7 to -3.1]
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant; Week 12: Total Symptom Score; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 13, analysis 1]; LSMean Difference = -6.3, 95% CI 2-sided [-9.9 to -2.8]

14. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) at Weeks 4, 8 and 12
Description: The SDS was a composite of 3 self-rated items designed to measure the extent to which 3 major sectors in a participant's life are impaired by panic, anxiety, phobic, or depressive symptoms. The participant rates the extent to which his/her 1- work/school, 2- social life, and 3- family life are impaired by his/her symptoms on a 10-point visual analog scale. The 3 items could be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired).Higher scores indicate significant functional impairment.
Time Frame: Baseline and weeks 4, 8 and 12
Population: ITT population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 42 | 40
score on a scale
  Week 4: Work/School: number analyzed (Participants) | 35 | 38
  Week 4: Work/School | -1.3 (2.43) | -3.6 (2.78)
  Week 8: Work/School: number analyzed (Participants) | 34 | 35
  Week 8: Work/School | -1.7 (2.56) | -4.4 (2.43)
  Week 12: Work/School: number analyzed (Participants) | 35 | 36
  Week 12: Work/School | -1.8 (2.76) | -4.3 (2.47)
  Week 4: Social Life | -1.2 (2.35) | -3.3 (2.60)
  Week 8: Social Life: number analyzed (Participants) | 39 | 40
  Week 8: Social Life | -1.3 (2.57) | -3.8 (2.79)
  Week 12: Social Life: number analyzed (Participants) | 40 | 40
  Week 12: Social Life | -1.5 (2.55) | -3.6 (2.51)
  Week 4: Family Life/Home Responsibilities | -1.5 (2.70) | -3.3 (2.97)
  Week 8: Family Life/Home Responsibilities: number analyzed (Participants) | 39 | 40
  Week 8: Family Life/Home Responsibilities | -1.7 (2.64) | -4.0 (2.83)
  Week 12: Family Life/Home Responsibilities: number analyzed (Participants) | 40 | 40
  Week 12: Family Life/Home Responsibilities | -1.7 (2.38) | -3.7 (2.65)
  Week 4: Global Functional Impairment: number analyzed (Participants) | 35 | 38
  Week 4: Global Functional Impairment | -3.7 (5.50) | -9.6 (6.99)
  Week 8: Global Functional Impairment: number analyzed (Participants) | 34 | 35
  Week 8: Global Functional Impairment | -4.5 (6.87) | -12.3 (6.42)
  Week 12: Global Functional Impairment: number analyzed (Participants) | 35 | 36
  Week 12: Global Functional Impairment | -4.8 (6.49) | -11.8 (6.35)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant; Week 4: Work/School; Test type: Superiority; p < 0.001, ANCOVA — Least square mean difference versus placebo, obtained from an ANCOVA model with treatment group as fixed effect and baseline SDS as covariate; LSMean Difference = -1.7, 95% CI 2-sided [-2.7 to -0.8]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant; Week 8: Work/School; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LSMean Difference = -2.0, 95% CI 2-sided [-2.8 to -1.3]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant; Week 12: Work/School; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LSMean Difference = -1.6, 95% CI 2-sided [-2.5 to -0.8]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant; Week 4: Social Life; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LSMean Difference = -1.4, 95% CI 2-sided [-2.2 to -0.6]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant; Week 8: Social Life; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LSMean Difference = -1.9, 95% CI 2-sided [-2.7 to -1.1]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant; Week 12: Social Life; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LSMean Difference = -1.6, 95% CI 2-sided [-2.4 to -0.7]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant; Week 4: Family Life/Home Responsibilities; Test type: Superiority; p = 0.005, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LSMean Difference = -1.3, 95% CI 2-sided [-2.2 to -0.4]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant; Week 8: Family Life/Home Responsibilities; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LSMean Difference = -1.7, 95% CI 2-sided [-2.5 to -0.9]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant; Week 12: Family Life/Home Responsibilities; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LSMean Difference = -1.6, 95% CI 2-sided [-2.4 to -0.7]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant; Week 4: Global Functional Impairment; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LSMean Difference = -4.4, 95% CI 2-sided [-6.9 to -2.0]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant; Week 8: Global Functional Impairment; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LSMean Difference = -5.8, 95% CI 2-sided [-8.0 to -3.6]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant; Week 12: Global Functional Impairment; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LSMean Difference = -5.3, 95% CI 2-sided [-7.8 to -2.8]

15. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) at Weeks 4, 8 and 12 (Days Lost and Days Unproductive)
Description: The SDS was a composite of 3 self-rated items designed to measure the extent to which 3 major sectors in a participant's life are impaired by panic, anxiety, phobic, or depressive symptoms. The participant rates the extent to which his/her 1- work/school, 2- social life, and 3- family life are impaired by his/her symptoms. In addition to the 3 items, the participants were asked two questions Days Lost: On how many days in the last week did your symptoms cause you to miss school or work or leave you unable to carry out your normal daily responsibilities? Day Unproductive: On how many days in the last week did you feel so impaired by your symptoms, that even though you went to school or work, your productivity was reduced?
Time Frame: Baseline and weeks 4, 8 and 12
Population: ITT population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 29 | 28
days
  Week 4: Days Lost: number analyzed (Participants) | 27 | 25
  Week 4: Days Lost | -0.2 (1.27) | 0.0 (0.73)
  Week 8: Days Lost: number analyzed (Participants) | 29 | 27
  Week 8: Days Lost | -0.3 (0.81) | 0.0 (0.00)
  Week 12: Days Lost: number analyzed (Participants) | 26 | 27
  Week 12: Days Lost | -0.2 (1.18) | 0.0 (0.00)
  Week 4: Days Unproductive: number analyzed (Participants) | 27 | 26
  Week 4: Days Unproductive | -0.8 (2.83) | -1.7 (2.67)
  Week 8: Days Unproductive | -1.2 (3.10) | -2.0 (2.55)
  Week 12: Days Unproductive: number analyzed (Participants) | 26 | 28
  Week 12: Days Unproductive | -1.4 (2.82) | -2.2 (2.59)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant; Week 4: Days Lost; Test type: Superiority; p = 0.936, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LSMean difference = 0.00, 95% CI 2-sided [-0.5 to 0.6]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant; Week 8: Days Lost; Test type: Superiority; p = 0.884, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LSMean difference = 0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant; Week 12: Days Lost; Test type: Superiority; p = 0.124, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.4 to 0.1]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant; Week 4: Days Unproductive; Test type: Superiority; p = 0.052, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-1.8 to 0.0]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant; Week 8: Days Unproductive; Test type: Superiority; p = 0.060, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LSMean difference = -0.9, 95% CI [-1.7 to 0.0]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant; Week 12: Days Unproductive; Test type: Superiority; p = 0.049, ANCOVA — [p-value comment as in outcome 14, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.7 to 0.0]

16. Secondary Outcome: Change From Baseline in Plasma Concentration of Luteinizing Hormone (LH)
Description: Change From baseline in plasma concentration of LH was reported.
Time Frame: Baseline and week 4: pre-dose, week 8:pre-dose, week 12:pre-dose, week 12: 3h, follow-up (week 15)
Population: Safety population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: international unit per liter (IU/L)
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 43 | 42
international unit per liter (IU/L)
  Week 4: Pre-dose | -2.34 (9.350) | -8.84 (10.865)
  Week 8: Pre-dose: number analyzed (Participants) | 40 | 40
  Week 8: Pre-dose | -3.86 (9.838) | -9.46 (13.647)
  Week 12: Pre-dose: number analyzed (Participants) | 40 | 40
  Week 12: Pre-dose | -4.61 (13.304) | -9.72 (12.834)
  Week 12: 3 hours (h): number analyzed (Participants) | 40 | 40
  Week 12: 3 hours (h) | -7.16 (13.009) | -21.78 (11.923)
  Week 15 | -6.16 (14.197) | -3.33 (11.742)

17. Secondary Outcome: Change From Baseline in Plasma Concentration of Follicle-Stimulating Hormone (FSH)
Description: Change From baseline in plasma concentration of FSH was reported.
Time Frame: Baseline and week 4: pre-dose, week 8:pre-dose, week 12:pre-dose, week 12:3h, follow-up (week 15)
Population: Safety population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 43 | 42
IU/L
  Week 4: Pre-dose: number analyzed (Participants) | 43 | 41
  Week 4: Pre-dose | -5.80 (19.430) | -3.44 (18.026)
  Week 8: Pre-dose: number analyzed (Participants) | 40 | 40
  Week 8: Pre-dose | -6.60 (20.086) | -10.36 (23.943)
  Week 12: Pre-dose: number analyzed (Participants) | 40 | 40
  Week 12: Pre-dose | -7.05 (19.978) | -10.51 (24.521)
  Week 12: 3h: number analyzed (Participants) | 40 | 40
  Week 12: 3h | -8.47 (19.159) | -19.48 (22.734)
  Week 15 | -6.50 (21.011) | -6.97 (22.273)

18. Secondary Outcome: Change From Baseline in Plasma Concentration of Estradiol (E2)
Description: Change From baseline in plasma concentration of E2 was reported.
Time Frame: Baseline and week 4: pre-dose, week 8:pre-dose, week 12:pre-dose, week 12:3h, follow-up (week 15)
Population: Safety population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: Picomoles per liter (pmol/L)
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 43 | 42
Picomoles per liter (pmol/L)
  Week 4: Pre-dose | 18.4 (140.36) | -7.3 (75.13)
  Week 8: Pre-dose: number analyzed (Participants) | 40 | 40
  Week 8: Pre-dose | 26.0 (157.18) | 1.0 (71.78)
  Week 12: Pre-dose: number analyzed (Participants) | 40 | 40
  Week 12: Pre-dose | 32.3 (101.87) | 25.5 (108.27)
  Week 12: 3h: number analyzed (Participants) | 40 | 40
  Week 12: 3h | 26.0 (100.33) | 11.5 (77.68)
  Week 15 | 37.0 (167.37) | 27.9 (188.18)

19. Secondary Outcome: Change From Baseline in Plasma Concentration of Sex Hormone-Binding Globulin (SHBG)
Description: Change From baseline in plasma concentration of SHBG was reported.
Time Frame: Baseline and week 4: pre-dose, week 8:pre-dose, week 12:pre-dose, week 12:3h, follow-up (week 15)
Population: Safety population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: Nanomoles per liter (nmol/L)
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 43 | 42
Nanomoles per liter (nmol/L)
  Week 4: Pre-dose: number analyzed (Participants) | 43 | 41
  Week 4: Pre-dose | 0.61 (16.260) | -0.47 (11.986)
  Week 8: Pre-dose: number analyzed (Participants) | 40 | 40
  Week 8: Pre-dose | 5.10 (20.713) | -1.37 (12.186)
  Week 12: Pre-dose: number analyzed (Participants) | 40 | 40
  Week 12: Pre-dose | 1.75 (18.090) | 0.36 (15.165)
  Week 12: 3h: number analyzed (Participants) | 40 | 40
  Week 12: 3h | 1.56 (18.658) | -1.49 (16.406)
  Week 15 | 1.92 (16.341) | -0.86 (13.540)

20. Secondary Outcome: Change From Baseline in Plasma Concentration of Leptin
Description: Change From baseline in plasma concentration of leptin was reported.
Time Frame: Baseline and week 4: pre-dose, week 8:pre-dose, week 12:pre-dose, week 12:3h, follow-up (week 15)
Population: Safety population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: nanogram per liter (ng/mL)
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 43 | 42
nanogram per liter (ng/mL)
  Week 4: Pre-dose: number analyzed (Participants) | 42 | 40
  Week 4: Pre-dose | 1.2436 (5.6269) | -2.2185 (6.9522)
  Week 8: Pre-dose: number analyzed (Participants) | 40 | 40
  Week 8: Pre-dose | 1.6225 (7.5029) | -1.7090 (6.9716)
  Week 12: Pre-dose: number analyzed (Participants) | 40 | 40
  Week 12: Pre-dose | 0.9668 (5.4301) | -0.4183 (11.0737)
  Week 12: 3h: number analyzed (Participants) | 40 | 40
  Week 12: 3h | -2.0755 (5.3193) | -4.2085 (8.5335)
  Week 15 | -0.9914 (14.6660) | -0.6031 (8.2519)

21. Secondary Outcome: Change From Baseline in Plasma Concentration of Insulin
Description: Change From baseline in plasma concentration of insulin was reported.
Time Frame: Baseline and week 4: pre-dose, week 8:pre-dose, week 12:pre-dose, week 12:3h, follow-up (week 15)
Population: Safety population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: micro units per milliliter (μU/mL)
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 43 | 42
micro units per milliliter (μU/mL)
  Week 4: Pre-dose: number analyzed (Participants) | 43 | 41
  Week 4: Pre-dose | -0.2767 (3.0971) | -0.7512 (3.8798)
  Week 8: Pre-dose: number analyzed (Participants) | 40 | 40
  Week 8: Pre-dose | 0.3525 (4.0903) | -0.5325 (3.6121)
  Week 12: Pre-dose: number analyzed (Participants) | 40 | 40
  Week 12: Pre-dose | -0.0825 (3.1593) | 0.1300 (4.7942)
  Week 12: 3h: number analyzed (Participants) | 40 | 40
  Week 12: 3h | 16.3225 (19.0210) | 14.4950 (19.2787)
  Week 15 | 0.3256 (4.1132) | -0.1595 (3.1071)

22. Secondary Outcome: Change From Baseline in Plasma Concentration of C-peptide
Description: Change From baseline in plasma concentration of C-peptide was reported.
Time Frame: Baseline and week 4: pre-dose, week 8:pre-dose, week 12:pre-dose, week 12:3h, follow-up (week 15)
Population: Safety population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 43 | 42
ng/mL
  Week 4: Pre-dose: number analyzed (Participants) | 43 | 41
  Week 4: Pre-dose | -0.0465 (0.3978) | -0.1463 (0.5134)
  Week 8: Pre-dose: number analyzed (Participants) | 40 | 40
  Week 8: Pre-dose | -0.0300 (0.5273) | -0.1175 (0.4750)
  Week 12: Pre-dose: number analyzed (Participants) | 40 | 40
  Week 12: Pre-dose | -0.0750 (0.5212) | -0.0425 (0.7154)
  Week 12: 3h: number analyzed (Participants) | 40 | 40
  Week 12: 3h | 2.1325 (1.9976) | 2.2875 (2.1811)
  Week 15 | -0.0047 (0.6102) | -0.0095 (0.4023)

23. Secondary Outcome: Change From Baseline in Plasma Concentration of Glycated Hemoglobin (HBA1c)
Description: Change From baseline in plasma concentration of HBA1C was reported.
Time Frame: Baseline and week 12
Population: Safety population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: Percentage of HBA1c
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 40 | 39
Percentage of HBA1c | -0.00050000 (0.003162278) | -0.002307692 (0.004845800)

24. Secondary Outcome: Number of Participants With Adverse Events (AE's)
Description: An AE is any untoward medical occurrence in a participant administered a study drug, & which does not necessarily have to have a causal relationship with treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with use of a medicinal product (mp) whether or not considered related to the mp. An AE is considered "serious" if it results in death, is life-threatening, results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, results in congenital anomaly or birth defect, requires inparticipant hospitalization or leads to prolongation of hospitalization, hospitalization for treatment/observation/examination caused by AE is to be considered as serious, discontinuation due to increases in liver enzymes, other medically important events. TEAE was defined as an AE observed from first dose date up to end of study.
Time Frame: From first dose of study drug until end of the study (Up to week 15)
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 44 | 43
participants
  At least one TEAE | 35 | 29
  At least one serious TEAE | 1 | 0
  At least one TEAE leading to death | 0 | 0
  At least one severe TEAE | 0 | 0
  At least one TEAE for which the study treatment was permanently stopped | 0 | 2
  At least one TEAE that was considered treatment related | 11 | 13

25. Secondary Outcome: Change From Baseline in Plasma Concentration of Bone Alkaline Phosphatase (BALP) at Week 12
Description: Change from baseline in plasma concentration of BALP was reported.
Time Frame: Baseline and week 12
Population: ITT population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (ug/mL)
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 40 | 40
microgram per milliliter (ug/mL) | 2.9 (5.43) | 1.7 (3.19)

26. Secondary Outcome: Change From Baseline in Plasma Concentration of Carboxy-terminal Telopeptide of Type I Collagen (CTX) at Week 12
Description: Change from baseline in plasma concentration of CTX was reported.
Time Frame: Baseline and week 12
Population: ITT population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Placebo | Fezolinetant
Number analyzed (Participants) | 40 | 40
ug/mL | -0.021 (0.1278) | 0.001 (0.1356)

ADVERSE EVENTS:
Time Frame: From first dose of study drug until end of the study (Up to week 15)
Arm/Group | Placebo | Fezolinetant
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/43
Serious Adverse Events (participants affected / at risk) | 1/44 | 0/43
Other Adverse Events (participants affected / at risk) | 18/44 | 18/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=44) | Fezolinetant (N=43)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=44) | Fezolinetant (N=43)
Palpitations (Cardiac disorders) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 3 (3)
Influenza (Infections and infestations) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 6 (10) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (1):
  • Study Protocol (2015-12-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT05419908/Prot_000.pdf